CLINICAL TRIAL: NCT06101758
Title: Prospective Study of Ultrasound Assessment of Sarcopenia and Correlated Clinical Outcomes in Patients With Chronic Liver Disease: the SARCOLIVER Study
Brief Title: Ultrasound Assessment of Sarcopenia in Patients With Chronic Liver Disease: the SARCOLIVER Study
Acronym: SARCOLIVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5855
Record Dates: First submitted 2023-09-04; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Liver Cirrhosis; Non-Alcoholic Fatty Liver Disease; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscular ultrasound assessment (Experimental): Adult patients aged 18-69 years with a diagnosis of either liver cirrhosis, non-alcoholic fatty liver disease or hepatocellular carcinoma
  Interventions: Diagnostic Test: Handgrip strength test; Diagnostic Test: total body Dual Energy X-Ray Absorptiometry (DXA); Diagnostic Test: Muscle ultrasound

INTERVENTIONS:
Diagnostic Test: Handgrip strength test — A handgrip strength test using a hydraulic hand dynamometer will be performed
Diagnostic Test: total body Dual Energy X-Ray Absorptiometry (DXA) — A total body Dual Energy X-Ray Absorptiometry (DXA) to estimate muscle mass will be performed
Diagnostic Test: Muscle ultrasound — A muscular ultrasound of abdominal muscles, forearm muscles, quadriceps and gastrocnemius will be performed

SUMMARY:
Sarcopenia is a complex multifactorial syndrome which could be present in older age (primary sarcopenia) or earlier in chronic disease (secondary sarcopenia). Even if in patients with chronic liver disease an association among sarcopenia and poor clinical outcomes is well known, the data available about the prevalence of sarcopenia in patients with liver cirrhosis, non-alcoholic fatty liver disease and hepatocellular carcinoma are very variable according to the populations in object and, furthermore, few data are available regarding the use of muscular ultrasound to detect this condition. The aim of this study is to define the prevalence of sarcopenia in patients with liver cirrhosis, non-alcoholic fatty liver disease and hepatocellular carcinoma in follow-up at our center and the clinical outcomes associated with this condition, and to determine the reliability of muscular ultrasound to diagnose the condition of sarcopenia through a comparison with other validated techniques such as computed tomography, magnetic resonance imaging and dual-energy X-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Ability to express informed consent
* Diagnosis of liver cirrhosis or non-alcoholic fatty liver disease or hepatocellular carcinoma based on clinical characteristics, biochemical serum tests and liver imaging examination or liver histologic examination if available

Exclusion Criteria:

* inability to express informed consent
* pregnancy
* presence of a concomitant oncologic disease different from hepatocellular carcinoma
* presence of a concomitant gastrointestinal disease able to influence the absorption and digestion of nutrients (e.g. inflammatory bowel disease, celiac disease, short-bowel syndrome, congenital defects of metabolism)
* presence of a concomitant gastrointestinal or neurologic disease able to influence the ability of feeding (e.g. dysphagia, parkinson disease, neuromuscular diseases, diseases of the autonomic nervous system, cognitive impairment or dementia)
* chronic kidney disease from stage 3 B (IIIB) according to Kidney Disease: Improving Global Outcomes (KDIGO) classification (eGFR <45ml/min/1.73m2)
* chronic heart failure from stage Ney York Heart Association (NYHA) II
* concomitant infection from Mycobacterium Tuberculosis or human immunodeficiency virus or chronic parasitic infections

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To calculate the prevalence of the condition of sarcopenia in patients with liver cirrhosis, non-alcoholic fatty liver disease and hepatocellular carcinoma | 24 months

SECONDARY OUTCOMES:
Association among sarcopenia and survival or acute decompensation events in patients with liver cirrhosis | 24 months
To calculate the prevalence of obesity with sarcopenia in patients with non-alcoholic fatty liver disease | 24 months
To evaluate the association among sarcopenia and therapeutic response in patients with hepatocellular carcinoma | 24 months
To calculate cohen's Kappa to evaluate the concordance among muscular ultrasound and dual-energy X-ray absorption, computed tomography scan and magnetic resonance imaging in the detection of sarcopenia | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CEMAD, Roma, RM, Italy